CLINICAL TRIAL: NCT01451541
Title: A 12-Week Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Safety and Efficacy Study of Ciclesonide Nasal Aerosol in Subjects 6-11 Years With Perennial Allergic Rhinitis
Brief Title: A Safety and Efficacy Study of Ciclesonide Nasal Aerosol in Subjects 6-11 Years With Perennial Allergic Rhinitis (PAR).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP060-306
Record Dates: First submitted 2011-10-11; First posted 2011-10-13 (Estimated); Results first posted 2014-05-06 (Estimated); Last update posted 2014-05-06 (Estimated); Status verified 2014-04

CONDITIONS: Perennial Allergic Rhinitis; PAR
MeSH Terms: conditions — Rhinitis, Allergic, Perennial

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- ciclesonide nasal aerosol 37mcg (Active Comparator): ciclesonide nasal aerosol 37mcg - the dose is administered as 1 actuation per nostril to give a total dose of 37mcg once daily
  Interventions: Drug: Ciclesonide nasal aerosol 37 mcg
- ciclesonide nasal aerosol 74 mcg (Active Comparator): ciclesonide nasal aerosol 74 mcg - the dose is administered as 1 actuation per nostril to give a total dose of 74 mcg once daily
  Interventions: Drug: ciclesonide nasal aerosol 74 mcg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ciclesonide nasal aerosol 37 mcg — ciclesonide nasal aerosol 37mcg - the dose is administered as 1 actuation per nostril to give a total dose of 37
  Arms: ciclesonide nasal aerosol 37mcg
Drug: ciclesonide nasal aerosol 74 mcg — ciclesonide nasal aerosol 74 mcg - the dose is administered as 1 actuation per nostril to give a total dose of 74 mcg
  Arms: ciclesonide nasal aerosol 74 mcg
Drug: Placebo — Placebo - one dose per nostril
  Arms: Placebo

SUMMARY:
This is a 12-week, multicenter, randomized, double-blind, placebo-controlled, parallel-group, efficacy and safety study of ciclesonide nasal aerosol administered once daily to male and premenarchal female subjects 6 to 11 years of age with a diagnosis of PAR.

DETAILED DESCRIPTION:
This is a 12-week, multicenter, randomized, double-blind, placebo-controlled, parallel-group, efficacy and safety study of ciclesonide nasal aerosol administered once daily to male and premenarchal female subjects 6 to 11 years of age with a diagnosis of PAR. This study will consist of the following periods/visits: Screening , Single-blind Placebo Run-in period, Double-blind Treatment period , Follow-up. The total duration of subject participation will be approximately 5 months.

ELIGIBILITY:
Inclusion Criteria:

* Gives written informed consent (parent/legal guardian) and assent (from the child), including privacy authorization as well as adherence to concomitant medication withholding periods, prior to participation.
* Is a male or premenarchal female 6 to 11 years old at the screening visit.
* Is in general good health (defined as the absence of any clinically relevant abnormalities as determined by the investigator) based on screening physical examination and medical history.
* Has a history of PAR to a relevant perennial allergen (house dust mites, cockroaches, molds, and animal dander) for a minimum of 1 year immediately preceding the study screening visit. The PAR must have been of sufficient severity to have required treatment (either continuous or intermittent) in the past and require treatment throughout the entire study period.
* Has a demonstrated sensitivity to at least 1 allergen known to induce PAR (house dust mites, cockroaches, molds, and animal dander) based on a documented result with a standard skin-prick test either within 12 months prior to screening visit or performed at the screening visit. A positive test is defined as a wheal diameter at least 3 mm larger than the negative control wheal for the skin-prick test. The subject's positive allergen test must be consistent with the medical history of PAR, and the allergen must be present in the subject's environment throughout the study.
* Subject or parent/guardian must possess an educational level and degree of understanding of English that enables them to communicate suitably with the Investigator and study coordinator as well as accurately complete both the AR diary and PRQLQ

Exclusion Criteria:

* Has a history of physical findings of nasal pathology, including nasal polyps or other clinically significant respiratory tract malformations; recent unhealed nasal biopsy; nasal trauma; or nasal ulcers or perforations. Surgery and atrophic rhinitis or rhinitis medicamentosa are not permitted within the 120 days prior to the screening visit.
* Has evidence of infection, significant anatomic abnormality, ulceration of the mucosa, blood in the nose, or any other clinically relevant finding on nasal examination at the screening visit.
* Has nasal jewelry.
* Has participated in any investigational drug trial within the 30 days preceding the screening visit or is planning participation in another investigational drug trial at any time during this trial.
* Has a known hypersensitivity to any corticosteroid or any of the excipients in the formulation of ciclesonide.
* Has a history of a respiratory infection or disorder, including but not limited to bronchitis, pneumonia, influenza, and severe acute respiratory syndrome, within the 14 days preceding the screening visit.
* Has active asthma requiring treatment with inhaled or systemic corticosteroids and/or routine use of beta-agonists and any controller drugs (eg, theophylline, leukotriene antagonists); intermittent use (≤ 3 uses per week) of inhaled short-acting beta-agonists is acceptable. Use of short-acting beta-agonists for exercise-induced bronchospasm will be allowed.
* Is expecting to use any disallowed concomitant medications during the treatment period.
* Is, in the investigator's judgment, having a seasonal exacerbation at the time of the screening visit or is likely to have one during the study.
* Is planning initiation of immunotherapy during the study period or dose escalation during the study period. However, initiation of immunotherapy 90 days or more prior to the screening visit and use of a stable (maintenance) dose (30 days or more) may be considered for inclusion.
* Has nonvaccinated exposure to or active infection with chickenpox or measles within the 21 days preceding the screening visit.
* Initiates pimecrolimus cream 1% or greater or tacrolimus ointment 0.03% or greater during the study period or plans a dose escalation during the study period. However, initiation of these creams/ointments 30 days or more prior to screening and use of a stable (maintenance) dose during the study period may be considered for inclusion.
* Is a child or relative of any clinical investigator or site personnel, even those who are not directly involved in this study.
* Resides in the same household as another subject who is participating in this study.
* Has any of the following conditions that are judged by the investigator to be clinically significant and/or to affect the subject's ability to participate in the clinical trial:

  * impaired hepatic function
  * history of ocular disturbances, eg, glaucoma or posterior subcapsular cataracts or herpes simplex
  * any systemic infection
  * hematological (including anemia), hepatic, renal, endocrine disease
  * gastrointestinal disease
  * malignancy (excluding basal cell carcinoma)
  * current neuropsychological condition with or without drug therapy. Any behavioral condition that could affect the subject's ability to accurately report symptoms to the caregiver such as developmental delay, attention deficit disorder, and autism.
* Has any condition that, in the judgment of the investigator, would preclude the subject from completing the protocol with the capture of the assessments as written.
* Has received ciclesonide nasal aerosol in a previous clinical trial.

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 848 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Respiratory Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (59):
- United States (59):
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Arkansas Pediatric Clinic, Little Rock, Arkansas
  - West Coast Clinical Trials, LLC, Costa Mesa, California
  - Premier Health Research Center, Downey, California
  - Allergy and Asthma Specialists Medical Group, Huntington Beach, California
  - Pediatric Care Medical Group, Huntington Beach, California
  - Allergy and Asthma Assoc of Southern CA, Mission Veijo, California
  - Center for Clinical Trials, LLC, Paramount, California
  - Allergy Associates Medical Group, San Diego, California
  - Allergy and Asthma Medical Group & Research Center, San Diego, California
  - Sansum Clinic, Santa Barbara, California
  - Colorado Allergy and Asthma Centers, PC, Centennial, Colorado
  - IMMUNOe International Research Centers, Centennial, Colorado
  - Storms Clinical Research Institute, Colorado Springs, Colorado
  - Ashtma and Allergy Associates, Pueblo, Colorado
  - DataQuest Medical Research, LLC, Lawerenceville, Georgia
  - Aeroallergy Research Labs of Savannah, Savannah, Georgia
  - Atlanta Allergy and Asthma Clinic, Stockbridge, Georgia
  - Clinical Research Atlanta, Stockton, Georgia
  - Sneeze, Wheeze, & Itch Associates, LLC, Normal, Illinois
  - College Park Family Care Center, Lenexa, Kansas
  - Family Allergy and Asthma Research Institute, Louisville, Kentucky
  - Gordon Raphael, MD, Bethesda, Maryland
  - Northeast Medical Research Associates Inc, North Dartmouth, Massachusetts
  - Respiratory Medicine Research Institute of Michigan, PLC, Ypsilanti, Michigan
  - Clinical Research Institute Inc, Plymouth, Minnesota
  - Clinical Research of the Ozarks, Warrensburg, Missouri
  - Clinical Research Group of Montana, Bozeman, Montana
  - The Asthma and Allergy Center, PC, Bellevue, Nebraska
  - Boys Town National Research Hospital, Boys Town, Nebraska
  - Atlantic Research Center LLC, Ocean City, New Jersey
  - Island Medical Research P.C., Rockville Centre, New York
  - Allergy and Asthma Center of NC, PA, High Point, North Carolina
  - Catalyst Medical Center, Fargo, North Dakota
  - Sterling Research Group Ltd, Cincinnati, Ohio
  - Toledo Center for Clinical Research, Sylvania, Ohio
  - Allergy, Asthma & Clinical Research Center, Oklahoma City, Oklahoma
  - Amy Darter, MD, Oklahoma City, Oklahoma
  - Cyn3rgy Research, Gresham, Oregon
  - Baker Allergy Asthma and Dermatolgy Research Center, LLC, Lake Oswego, Oregon
  - Clinical Research Institute of Southern Oregon, PC, Medford, Oregon
  - Allergy Associates Research Center, Portland, Oregon
  - Valley Clinical Research Center, Bethlehem, Pennsylvania
  - Asthma and Allergy Research Associates, Upland, Pennsylvania
  - National Allergy, Ashtma, and Urticaria Centers of Charleston, PA, North Charleston, South Carolina
  - Isis Clinical Research LLC, Austin, Texas
  - Sirius Clinical Research, Austin, Texas
  - TTS Research, Boerne, Texas
  - Pharmaceutical Research and Consulting, Inc., Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Kerrville Research Associates, Kerrville, Texas
  - Central Texas Health Research, New Braunfels, Texas
  - Sylvana Research Associates, San Antonio, Texas
  - Allergy and Asthma Research Institute, Waco, Texas
  - J. Lewis Research Inc., Salt Lake City, Utah
  - J. Lewis Research Inc., South Jordan, Utah
  - PI-Coor Clinical Research, Burke, Virginia
  - Clinical Research Partners, LLC, Henrico, Virginia
  - ASTHMA, Inc., Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Started | 283 | 282 | 281 (283 randomized. ITT = 281 (2 subjects discontinued prior to study medication).)
Completed | 247 | 257 | 254
Not Completed | 36 | 25 | 27
Not completed — Adverse Event | 4 | 3 | 6
Not completed — Lack of Efficacy | 2 | 0 | 0
Not completed — Lost to Follow-up | 4 | 4 | 7
Not completed — Withdrawal by Subject | 15 | 8 | 6
Not completed — randomization error, noncompliance | 11 | 10 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg | Total
Number analyzed (Participants) | 283 | 282 | 281 | 846
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 283 | 282 | 281 | 846
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 120 | 113 | 130 | 363
  Male | 163 | 169 | 151 | 483
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 1 | 3
  Asian | 5 | 2 | 7 | 14
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 37 | 43 | 39 | 119
  White | 224 | 216 | 216 | 656
  More than one race | 8 | 10 | 8 | 26
  Unknown or Not Reported | 9 | 9 | 9 | 27
Race/Ethnicity, Customized [Number; unit: participants]
  Hispanic or Latino | 89 | 101 | 91 | 281
  Unknown or Not Reported | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 194 | 181 | 190 | 565
Region of Enrollment [Number; unit: participants]
  United States | 283 | 282 | 281 | 846

OUTCOME MEASURES:

1. Primary Outcome: The Change From Baseline in Average Daily Subject-reported AM and PM Reflective Total Nasal Symptom Scores (rTNSS) Averaged Weekly Over the First 6 Weeks of the Double-blind Treatment.
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where: 0 = absent 1 = mild 2 = moderate 3 = severe Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. Difference was calculated as the six week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Weeks 0-6
Population: The Intent to Treat (ITT) population: All randomized subjects who received at least one dose of double blind study medication.Subjects with either missing baseline data or postdose data, or both and were not included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 278 | 280 | 275
units on a scale | -1.51 (0.130) | -2.10 (0.130) | -1.98 (0.131)
Statistical Analysis 1: Comparison: Placebo vs Ciclesonide Nasal Aerosol 37mcg; Using an estimate of the standard deviation of 2.2 for the change from baseline in daily average subject-reported AM and PM rTNSS averaged over the first 6 weeks of double-blind treatment, 284 subjects per treatment group would have provided 90% power to detect a mean difference between treatment groups of 0.6 in the change from baseline with a 2-sided significance level of 0.05. Approx. 852 subjects were randomly assigned in a 1:1:1 ratio (ie, approximately 284 subjects per treatment group); Test type: Superiority or Other; p < 0.05, Bonferroni-based gatekeeping method — Multiple comparisons were adjusted for the primary and key secondary endpoints; Bonferroni-based gatekeeping method was used for multiple comparison adjustment; LS Means with adjusted pvalues = 0.59
Statistical Analysis 2: Comparison: Placebo vs Ciclesonide Nasal Aerosol 74 mcg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Bonferroni-based gatekeeping method — Multiple comparisons were adjusted for the primary and key secondary endpoints; Bonferroni-based gatekeeping method was used for multiple comparison adjustment; LS Means with adjusted p-values. = 0.47

2. Secondary Outcome: Change From Baseline in Average Daily Subject-reported AM and PM Instantaneous Total Nasal Symptom Scores (iTNSS) Averaged Weekly Over the First 6 Weeks of Double-blind Treatment
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where: 0 = absent 1 = mild 2 = moderate 3 = severe Therefore, iTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TNSS measures these symptoms over the previous 10 minute time interval. Difference was calculated as the six week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Weeks 0 -6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 278 | 280 | 276
units on a scale | -1.29 (0.122) | -1.77 (0.122) | -1.72 (0.123)

3. Secondary Outcome: Change From Baseline in the Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) Overall Score at the End of the First 6 Weeks of Double-blind Treatment
Description: PRQLQ was developed to measure the functional problems (physical, emotional, and social) that are most troublesome to children with rhinoconjunctivitis. The PRQLQ has 23 questions in 5 domains (nose symptoms, eye symptoms, practical problems, activity limitation, and other symptoms). Children recalled how they were during the previous week and responded to each question on a 7-point scale (0 = not bothered to 6 = extremely bothered or 0 = none of the time to 6 = all of the time) for a total possible score of 138. The overall PRQLQ score is the mean of all 23 responses.
Time Frame: Weeks 0 -6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 269 | 268 | 270
units on a scale | -0.39 (0.05) | -0.51 (0.05) | -0.30 (0.054)

4. Secondary Outcome: Change From Baseline in Daily Average Subject-reported AM and PM rTNSS Averaged Weekly Over the 12-week Double-blind Treatment Period
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where: 0 = absent 1 = mild 2 = moderate 3 = severe Therefore, rTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Reflective TNSS measures these symptoms over the previous 12-hour time interval. Difference was calculated as the twelve week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement
Time Frame: Weeks 0 -12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 278 | 280 | 275
units on a scale | -1.92 (0.13) | -2.60 (0.14) | -2.47 (0.14)

5. Secondary Outcome: Change From Baseline in Daily Average Subject-reported AM and PM iTNSS Averaged Weekly Over the 12-week Double-blind Treatment Period
Description: TNSS is the sum of individual symptoms of runny nose, sneezing, itchy nose, and nasal congestions. Subjects assess each individual symptoms on a scale of 0-3 where: 0 = absent 1 = mild 2 = moderate 3 = severe Therefore, iTNSS values range from 0-12 (with 0 representing an absence of symptoms and higher scores reflecting more severe symptoms). Instantaneous TNSS measures these symptoms over the previous 10 minute time interval. Difference was calculated as the twelve week treatment average - baseline. Greater reductions in the change from baseline score indicate greater improvement.
Time Frame: Weeks 0 -12
Population: The Intent to Treat (ITT) population: All randomized subjects who received at least one dose of double blind study medication.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 278 | 280 | 276
units on a scale | -1.69 (0.13) | -2.22 (0.13) | -2.15 (0.13)

6. Secondary Outcome: Change From Baseline in Daily Average Subject-reported AM iTNSS Averaged Over the First 6 Weeks of Double-blind Treatment
Description: as for outcome 2
Time Frame: Weeks 0 -6
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 278 | 280 | 276
units on a scale | -1.26 (0.12) | -1.75 (0.12) | -1.74 (0.12)

7. Secondary Outcome: Change From Baseline in Daily PRQLQ Overall Score at the End of the 12-week Double-blind Treatment Period
Description: as for outcome 3
Time Frame: Weeks 0 -12
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 271 | 269 | 272
units on a scale | -0.54 (0.059) | -0.68 (0.059) | -0.47 (0.059)

8. Secondary Outcome: Time to Maximal Effect [Time to >= 90% Maximum Difference From Placebo in LS Means (Days)]
Description: The time to maximal effect is defined as the number of days until the first treatment day on which the estimated difference between active ciclesonide nasal aerosol and placebo is at least 90% of the largest estimated difference.This is based on the analyses of change from baseline in the average of AM and PM reflective TNSS scores for each day. The time to achieve at least 90% of these estimated differences was calculated.
Time Frame: Weeks 0 -6
Population: as for outcome 5
Measure: Number; unit: Number of Days
Arm/Group | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 282 | 281
Number of Days | 39 | 10

9. Secondary Outcome: Number of Subjects Experiencing AEs, SAEs, and Discontinuations Due to AEs
Time Frame: Weeks 0 -12
Measure: Number; unit: participants
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 283 | 282 | 281
participants
  Any TEAE | 154 | 142 | 143
  Any TEAE during first 6 weeks of double-blind | 114 | 99 | 102
  Potentially related AE | 46 | 39 | 46
  Local AE | 49 | 45 | 46
  Discontinued study drug due to an AE | 4 | 3 | 6
  Severe AE | 12 | 14 | 17
  Serious AE | 1 | 1 | 2

10. Secondary Outcome: Percentage of Subjects Experiencing AEs, SAEs, and Discontinuations Due to AEs
Time Frame: Weeks 0 -12
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 283 | 282 | 281
percentage of subjects
  Any TEAE | 54.4 | 50.4 | 50.9
  Any TEAE during first 6 weeks of double-blind | 40.3 | 35.1 | 36.3
  Potentially related AE | 16.3 | 13.8 | 16.4
  Local AE | 17.3 | 16.0 | 16.4
  Discontinued study drug due to an AE | 4 | 3 | 6
  Severe AE | 4.2 | 5.0 | 6.0
  Serious AE | 0.4 | 0.4 | 0.7

11. Secondary Outcome: Number of Subjects Experiencing Nasal AEs, Including Epistaxis, Nasal Ulceration, and Nasal Perforation
Time Frame: Weeks 0 -12
Measure: Number; unit: participants
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 283 | 282 | 281
participants
  ACUTE SINUSITIS | 1 | 2 | 1
  APPLICATION SITE PAIN | 3 | 3 | 1
  EPISTAXIS | 26 | 20 | 26
  FACE INJURY | 2 | 1 | 4
  INCREASED UPPER AIRWAY SECRETION | 1 | 0 | 0
  MUCOSAL DISCOLOURATION | 1 | 0 | 0
  MUCOSAL EXCORIATION | 0 | 1 | 0
  MUCOSAL HAEMORRHAGE | 0 | 0 | 1
  NASAL CONGESTION | 0 | 3 | 1
  NASAL DISCOMFORT | 6 | 4 | 8
  NASAL DRYNESS | 0 | 0 | 1
  NASAL MUCOSAL DISCOLOURATION | 0 | 1 | 0
  NASAL MUCOSAL DISORDER | 4 | 0 | 2
  NASAL OEDEMA | 4 | 3 | 3
  NASAL SEPTUM DISORDER | 0 | 1 | 1
  NASAL SEPTUM ULCERATION | 1 | 0 | 1
  NASAL TURBINATE ABNORMALITY | 1 | 1 | 2
  NASAL ULCER | 0 | 0 | 1
  POSTNASAL DRIP | 0 | 1 | 1
  RHINALGIA | 0 | 0 | 1
  RHINITIS PERENNIAL | 4 | 0 | 1
  RHINORRHOEA | 2 | 1 | 1
  SCAB | 1 | 0 | 2
  SCRATCH | 1 | 0 | 0
  SINUS HEADACHE | 0 | 1 | 1
  SINUSITIS | 5 | 6 | 4
  SNEEZING | 7 | 1 | 0

12. Secondary Outcome: Percentage of Subjects Experiencing Nasal AEs, Including Epistaxis, Nasal Ulceration, and Nasal Perforation
Time Frame: Weeks 0 -12
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Number analyzed (Participants) | 283 | 282 | 281
percentage of subjects
  ACUTE SINUSITIS | 0.4 | 0.7 | 0.4
  APPLICATION SITE PAIN | 1.1 | 1.1 | 0.4
  EPISTAXIS | 9.2 | 7.1 | 9.3
  FACE INJURY | 0.7 | 0.4 | 1.4
  INCREASED UPPER AIRWAY SECRETION | 0.4 | 0 | 0
  MUCOSAL DISCOLOURATION | 0.4 | 0 | 0
  MUCOSAL EXCORIATION | 0 | 0.4 | 0
  MUCOSAL HAEMORRHAGE | 0 | 0 | 0.4
  NASAL CONGESTION | 0 | 1.1 | 0.4
  NASAL DISCOMFORT | 2.1 | 1.4 | 2.8
  NASAL DRYNESS | 0 | 0 | 0.4
  NASAL MUCOSAL DISCOLOURATION | 0 | 0.4 | 0
  NASAL MUCOSAL DISORDER | 1.4 | 0 | 0.7
  NASAL OEDEMA | 1.4 | 1.1 | 1.1
  NASAL SEPTUM DISORDER | 0 | 0.4 | 0.4
  NASAL SEPTUM ULCERATION | 0.4 | 0 | 0.4
  NASAL TURBINATE ABNORMALITY | 0.4 | 0.4 | 0.7
  NASAL ULCER | 0 | 0 | 0.4
  POSTNASAL DRIP | 0 | 0.4 | 0.4
  RHINALGIA | 0 | 0 | 0.4
  RHINITIS PERENNIAL | 1.4 | 0 | 0.4
  RHINORRHOEA | 0.7 | 0.4 | 0.4
  SCAB | 0.4 | 0 | 0.7
  SCRATCH | 0.4 | 0 | 0
  SINUS HEADACHE | 0 | 0.4 | 0.4
  SINUSITIS | 1.8 | 2.1 | 1.4
  SNEEZING | 2.5 | 0.4 | 0

ADVERSE EVENTS:
Time Frame: 0-12 weeks
Arm/Group | Placebo | Ciclesonide Nasal Aerosol 37mcg | Ciclesonide Nasal Aerosol 74 mcg
Serious Adverse Events (participants affected / at risk) | 1/283 | 1/282 | 2/281
Other Adverse Events (participants affected / at risk) | 83/283 | 95/282 | 85/281
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=283) | Ciclesonide Nasal Aerosol 37mcg (N=282) | Ciclesonide Nasal Aerosol 74 mcg (N=281)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=283) | Ciclesonide Nasal Aerosol 37mcg (N=282) | Ciclesonide Nasal Aerosol 74 mcg (N=281)
PYREXIA (General disorders) | 12 (13) | 18 (20) | 17 (17)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 18 (20) | 24 (25) | 25 (29)
HEADACHE (Nervous system disorders) | 25 (42) | 31 (44) | 25 (38)
COUGH (Respiratory, thoracic and mediastinal disorders) | 19 (22) | 21 (25) | 15 (22)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 26 (42) | 20 (25) | 26 (45)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 17 (19) | 15 (16) | 10 (14)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish